CLINICAL TRIAL: NCT01572272
Title: Comparison of Open Versus Masked Distal EtCO2 Monitoring of Neonates Ventilated With Conventional Ventilation. A Randomized, Multi-Center Study
Brief Title: Comparison of Open Versus Masked Distal EtCO2 Monitoring of Neonates Ventilated With Conventional Ventilation
Status: Completed | Type: Observational
Sponsor: Oridion (Industry)
Responsible Party: Sponsor
Organization: Medtronic - MITG (Industry)
Other Study IDs: D007157
Record Dates: First submitted 2012-03-25; First posted 2012-04-06 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Intubated Neonates That Require Conventional Ventilation
Keywords: Distal Capnography; CO2; neonates; conventional ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Open: Open group: Data derived from the Capnostream20p and displayed to the medical team. It will allow the treating physician and the nursing team to review the real time data and make clinical decisions based upon it if felt necessary.
- Masked: Data derived from the Capnostream20p will be recorded; however the medical staff will be masked from it and hence will not use it.

SUMMARY:
Primary:

The purpose of this study is to assess the clinical implications of continuous distal CO2 monitoring when used for clinical decisions

Sub Study:

• Evaluate the average life time (duration) of Standard Carinal VitaLine set in comparison to the Carinal VitaLine set that its sampling tubing is made of PEBAX (dehumidifying material).

Description of Study Design:

Patients will be randomized at the baseline evaluation visit into one of the following groups:

* Masked group: Data derived from the Capnostream20p will be recorded; however the medical staff will be masked from it and hence will not use it.
* Open group: Data derived from the Capnostream20p and displayed to the medical team. It will allow the treating physician and the nursing team to review the real time data and make clinical decisions based upon it if felt necessary.

ELIGIBILITY:
Inclusion Criteria:

* Intubated neonates with double-lumen ETT (Uncuffed Tracheal Tube, Mallinckrodt Inc., Chih, Mexico) that their respiratory condition requires conventional ventilation.
* Obtaining signed Informed Consent Form by the parents or legal guardian
* Intubated neonates that are expected to provide at least 3 pairs of blood samples and ETCO2 measurements during ventilation period

Exclusion Criteria:

* Intubated neonates with single-lumen ETTs
* Neonates who are ventilated with HFV
* Any significant medical condition which, at the investigator's discretion, may interfere with the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Intubated neonates that require conventional ventilation
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2012-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Compare between the open and the masked group in the following: the percentage of measurement points at the Safe range: 60>PaCO2>30, Normal range 45>PaCO2>35 and Adequate (permissive) range: 45-55. | 2 weeks
  Participants will be follwed throughout the duration of the ventilation. Estimated time: 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Amir Kugelman, Prof., Principal Investigator — Bnai Zion MC, Haifa Israel
Locations (3):
- Israel (3):
  - Soroka MC, Beersheba
  - Bnai Zion MC, Haifa
  - Shaare Zedek MC, Jerusalem

REFERENCES:
- [Derived] Kugelman A, Golan A, Riskin A, Shoris I, Ronen M, Qumqam N, Bader D, Bromiker R. Impact of Continuous Capnography in Ventilated Neonates: A Randomized, Multicenter Study. J Pediatr. 2016 Jan;168:56-61.e2. doi: 10.1016/j.jpeds.2015.09.051. Epub 2015 Oct 17. PMID 26490126